CLINICAL TRIAL: NCT05747248
Title: Tracheal, Lung, and Diaphragmatic Ultrasonography Applications for Rapid Confirmation of Endotracheal Tube Position
Status: Completed | Type: Observational
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Islam Galal Sayed, Professor, Aswan University
Other Study IDs: ETT position confimation by US
Record Dates: First submitted 2023-02-17; First posted 2023-02-28 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Endotracheal Intubation
Keywords: ETT
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography — Tracheal, diaphragmatic and lung ultrasonography

SUMMARY:
Nowadays endotracheal intubation is considered a fundamental management procedure during emergency resuscitation. Unrecognized misplacement of the ETT during endotracheal intubation and ventilation, has a reported incidence of 2.9-16.7% and is a frequent cause of morbidity and mortality in emergency intubations. The aim of this study is to determine the diagnostic accuracy of the tracheal, diaphragmatic and sonographic estimation of lung sliding for the rapid verification of endotracheal tube position in the intensive care unit (RICU) with reference to Co₂ monitors (capnography) (the gold standard technique)

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old with endotracheal intubation
* Having normal airway anatomy

Exclusion Criteria:

* Age below 18 years old
* Neck deformities,
* Presence in history of neck radiation,
* Cervical spine immobility/instability
* Unstable vital signs
* Unwilling to participate or denial of informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients intubated with a cuff ETT
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-08-20 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
The verification of endotracheal tube position using the ultrasonography in the respiratory intensive care unit (RICU) with reference to Co₂ monitors (capnography) (the gold standard technique) | one hour
  The confirmation of endotracheal tube position using the tracheal, diaphragmatic and sonographic estimation of lung sliding for the rapid verification of endotracheal tube position in the intensive care unit (RICU) with reference to Co₂ monitors (capnography) (the gold standard technique)

CONTACTS AND LOCATIONS:
Locations (1):
- Islam Galal Sayed, Asyut, Egypt

REFERENCES:
- [Background] Sethi AK, Salhotra R, Chandra M, Mohta M, Bhatt S, Kayina CA. Confirmation of placement of endotracheal tube - A comparative observational pilot study of three ultrasound methods. J Anaesthesiol Clin Pharmacol. 2019 Jul-Sep;35(3):353-358. doi: 10.4103/joacp.JOACP_317_18. PMID 31543584